CLINICAL TRIAL: NCT01364259
Title: A Randomized, Placebo-controlled Trial of Amifostine for Prevention of Facial Numbness in Patients Receiving Stereotactic Radiosurgery for Trigeminal Neuralgia
Brief Title: A Study of Amifostine for Prevention of Facial Numbness in Radiosurgery Treatment of Trigeminal Neuralgia
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Patterns of practice changed and this technique is no longer used.
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Scott Soltys, Assistant Professor, Stanford University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB-14896; SU-05252011-7806 (Other: Stanford alternate number)
Record Dates: First submitted 2011-05-26; First posted 2011-06-02 (Estimated); Results first posted 2017-04-04 (Actual); Last update posted 2017-04-04 (Actual); Status verified 2017-02

CONDITIONS: Trigeminal Neuralgia
Keywords: tic douloureux
MeSH Terms: conditions — Trigeminal Neuralgia | interventions — Amifostine; Radiosurgery

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator): Placebo and SRS
  Interventions: Procedure: CyberKnife stereotactic radiosurgery
- Amifostine (Experimental): Amifostine and CyberKnife stereotactic radiosurgery
  Interventions: Drug: Amifostine

INTERVENTIONS:
Drug: Amifostine — Amifostine and CyberKnife stereotactic radiosurgery
  Other Names: CyberKnife stereotactic radiosurgery
  Arms: Amifostine
Procedure: CyberKnife stereotactic radiosurgery — CyberKnife stereotactic radiosurgery
  Arms: Placebo

SUMMARY:
Trigeminal neuralgia or tic douloureux is severe, often debilitating, facial pain that significantly impairs the patient's quality of life and health. Stereotactic radiosurgery has been shown to provide pain relief in majority of patients treated. However, a common side effect of radiosurgery is facial numbness. Our goal is to maximize pain control while minimizing side effects. To this end, the purpose of this study is to evaluate whether adding a drug, amifostine, at the time of radiosurgery will protect patients from facial numbness.

DETAILED DESCRIPTION:
Patients will be evaluated by a multi-disciplinary team composed of radiation oncologists and neurosurgeons. Pretreatment pain, neurologic function (including facial numbness), and health related quality of life will be assessed. Patients will be treated in a single session with 75 Gy maximal dose covering a 6 mm segment of the retrogasserian cisternal portion of the trigeminal sensory root. Treatment will be delivered using the CyberKnife Robotic Radiosurgery System with the patient in the supine position. An aquaplast head mask will be used to ensure adequate immobilization during therapy. The target volume shall be the 6 mm segment of the retrogasserian cisternal portion of the trigeminal sensory root. Patients will receive subcutaneous injection of amifostine (500 mg) or placebo 30 minutes +/- 30 minutes prior to SRS. Facial pain will be assessed using the Visual Analog Scale and Short-form McGill Pain Questionnaire. Following SRS, patients will be followed at 1, 3, 6, and 9 months ±7 days. Facial numbness will be assessed using the Barrow Neurologic Institute (BNI) Facial Numbness Score. Patient reported BNI facial numbness scoring and complete cranial nerve exam by a physician will be performed pre-treatment and at follow-up visits.

ELIGIBILITY:
Inclusion Criteria:

All patients age 18 years and older with typical trigeminal neuralgia, as determined by diagnostic criteria set by the International Headache Society, who are:

* Intolerant of or refractory to medical management; AND
* Not candidates for or refusing a surgical micro-vascular decompression.

Exclusion Criteria:

* Patients who present with pre-existing BNI grade III or IV facial numbness.
* Patients who have previously been treated with MVD.
* Patients who have previously had an ablative treatment, including prior SRS.
* Pediatric patients (age <18), pregnant women, and patients who are unable to give informed consent will be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2008-09; Primary Completion 2014-01 (Actual); Study Completion 2015-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clara Choi, Principal Investigator — Stanford University; Scott Soltys, Principal Investigator — Stanford University
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients will be evaluated by a multi-disciplinary team composed of radiation oncologists and neurosurgeons. During their visit, a physician or research coordinator will explain the study. Patients will be given the informed consent form to read. If they agree to participate, they will be asked to sign the consent form prior to participating.
Pre-assignment Details: Patient's pretreatment pain, neurologic function (including facial numbness), and health related quality of life will be assessed.
Groups:
- Placebo: Placebo and SRS
  CyberKnife stereotactic radiosurgery (srs)
- Amifostine: Amifostine and SRS
  CyberKnife stereotactic radiosurgery and Amifostine
Period: Overall Study
Arm/Group | Placebo | Amifostine
Started | 9 | 8
Completed | 9 | 8
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Placebo: Placebo and SRS
  CyberKnife stereotactic radiosurgery + saline
- Amifostine: Amifostine and CyberKnife stereotactic radiosurgery
  CyberKnife stereotactic radiosurgery + amofostine
- Total: Total of all reporting groups
Arm/Group | Placebo | Amifostine | Total
Number analyzed (Participants) | 9 | 8 | 17
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 1 | 1 | 2
  >=65 years | 8 | 7 | 15
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 7 | 12
  Male | 4 | 1 | 5
Region of Enrollment [Number; unit: participants]
  United States | 9 | 8 | 17

OUTCOME MEASURES:

1. Primary Outcome: Facial Numbness Following Radiosurgery
Description: Percent of patients with facial numbness following radiosurgery will be determined at one year follow up.
Time Frame: 1 year
Population: One subject randomized to drug arm did not have data.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Amifostine
Number analyzed (Participants) | 9 | 7
Participants | 7 | 6

2. Secondary Outcome: Pain Relief Following Radiosurgery
Description: Pain improvement as assessed by the Barrow Neurological Institute (BNI) facial pain score from pre-treatment baseline of BNI 3-5 (3-some pain/controlled on medications, 4-some pain/not controlled on medications, 5-severe pain) to BNI 1-2 (1-no pain/ no medication, 2- occasional pain/no medication)
Time Frame: 1 year
Population: 8 subjects were enrolled on the Amifostine arm, however, one subject was enrolled but withdrew prior to treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Amifostine
Number analyzed (Participants) | 9 | 7
Participants | 9 | 5
Statistical Analysis 1: Comparison: Placebo vs Amifostine; Test type: Superiority or Other; p = 0.175, Fisher Exact; Odds Ratio (OR) = 0 — Our odds ratio is equal to 0*5/9*2 because we have a zero cell in the two by two table. Hence the OR = 0

ADVERSE EVENTS:
Time Frame: Data was collected for 9 months.
Arm/Group | Placebo | Amifostine
Serious Adverse Events (participants affected / at risk) | 0/9 | 0/7
Other Adverse Events (participants affected / at risk) | 0/9 | 0/7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes